CLINICAL TRIAL: NCT04311554
Title: Aging With Dignity, Health, Optimism and Community
Acronym: ADHOC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mazonson & Santas Inc. (Industry)
Collaborators: Peter Shalit MD and Associates (Unknown); Red River Family Practice (Unknown); Central Texas Clinical Research (Unknown); Rosedale Infectious Diseases (Unknown); Midland Medical Center (Unknown); Anthony Mills MD Inc (Unknown); Stanford University (Other); Whitman-Walker Institute (Other Government); University of California, San Diego (Other); Ruth M. Rothstein CORE Center (Other); University of Wisconsin, Madison (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ADHOC-1001
Record Dates: First submitted 2020-03-02; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: HIV; PLWH; Aging; Older

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ADHOC is an observational study of people living with HIV over the age of 50. Data from this study will be used to research the interaction between HIV and aging.

DETAILED DESCRIPTION:
ADHOC is an observational study that collects data on PLWH over the age of 50 using an online questionnaire. The questionnaire includes information on sociodemographic factors, activities and interests, HIV diagnosis and status, health care use and satisfaction, antiretroviral therapy, comorbid medical conditions, health and well-being, substance use, and sexual practices.

ELIGIBILITY:
Eligibility criteria:

* have an HIV-1 or -2 infection,
* be ≥ 50 years of age,
* have no known acute medical problems requiring immediate inpatient treatment,
* be able to read and write in English, and
* be able and willing to provide online informed consent and complete the profile online.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People over the age of 50 with an HIV-1 or -2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 1049 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2022-10-19 (Estimated); Study Completion 2022-10-19 (Estimated)

PRIMARY OUTCOMES:
Change in loneliness | Through study completion, an average of 1 year
  Measured using the Three-Item Loneliness Scale. This scale is comprised of 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation.
Loneliness at baseline | Baseline
  Measured using the Three-Item Loneliness Scale. This scale is comprised of 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation.
Change in quality of life | Through study completion, an average of 1 year
  Measured using the PozQoL. PozQoL is a short 13-question scale assessing quality of life among people living with HIV. The scale includes four subscales: health concerns, psychological, social and functional.
Quality of life at baseline | Baseline
  Measured using the PozQoL. PozQoL is a short 13-question scale assessing quality of life among people living with HIV. The scale includes four subscales: health concerns, psychological, social and functional.
Change in cognitive function | Through study completion, an average of 1 year
  Measured using the Functional Assessment of HIV Infection (FAHI Cognition). The FAHI Cognition subscale will be used to create a standardized score to assess outcome.
Cognitive function at baseline | Baseline
  Measured using the Functional Assessment of HIV Infection (FAHI). The FAHI Cognition subscale will be used to create a standardized score to assess outcome.
Change in social well-being | Through study completion, an average of 1 year
  Measured using the Functional Assessment of HIV Infection (FAHI). The FAHI Social Well-being subscale will be used to create a standardized score to assess outcome.
Social well-being at baseline | Baseline
  Measured using the Functional Assessment of HIV Infection (FAHI). The FAHI Social Well-being subscale will be used to create a standardized score to assess outcome.
Change in depression | Through study completion, an average of 1 year
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Depression at baseline | Baseline
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Change in anxiety | Through study completion, an average of 1 year
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Anxiety at baseline | Baseline
  Measured using the Patient Health Questionnaire - 4 (PHQ-4). PHQ-4 is a brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Change in sleep quality | Through study completion, an average of 1 year
  Measured using The Medical Outcomes Study Sleep Scale (MOS-SS). MOS-SS includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache.
Sleep quality at baseline | Baseline
  Measured using The Medical Outcomes Study Sleep Scale (MOS-SS). MOS-SS includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache.
Change in alcohol use | Through study completion, an average of 1 year
  Measured using the Alcohol Use Disorder Identification Test (AUDIT-C). The AUDIT-C is a 3-item screening survey that can help identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence).
Alcohol use at baseline | Baseline
  Measured using the Alcohol Use Disorder Identification Test (AUDIT-C). The AUDIT-C is a 3-item screening survey that can help identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence).
Change in self-perceived stigma | Through study completion, an average of 1 year
  Measured using the Internalized AIDS-Related Stigma scale (IAS). IAS is a six-item scale designed to measure the construct of internalized stigma.
Self-perceived stigma at baseline | Baseline
  Measured using the Internalized AIDS-Related Stigma scale (IAS). IAS is a six-item scale designed to measure the construct of internalized stigma.
Change in lipodystrophy | Through study completion, an average of 1 year
  Measured using the Assessment of Body Change and Distress (ABCD). The ABCD assesses subjective report of bodily changes and body dissatisfaction, and it includes 20 items on the impact of bodily changes on psychosocial variables, quality of life, and HIV self-care behaviors.
Lipodystrophy at baseline | Baseline
  Measured using the Assessment of Body Change and Distress (ABCD). The ABCD assesses subjective report of bodily changes and body dissatisfaction, and it includes 20 items on the impact of bodily changes on psychosocial variables, quality of life, and HIV self-care behaviors.
Change in resilience | Through study completion, an average of 1 year
  Measured using the Connor-Davidson Resilience Scale (CD-RISC 2). The CD-RISC contains two items and was developed as a measure of "bounce-back" and adaptability.
Resilience at baseline | Baseline
  Measured using the Connor-Davidson Resilience Scale (CD-RISC 2). The CD-RISC contains two items and was developed as a measure of "bounce-back" and adaptability.
Change in interpersonal support | Through study completion, an average of 1 year
  Measured using the Interpersonal Support Evaluation Checklist - 6 (ISEL-6). ISEL-6 is derived from the long form of the ISEL and contains 6 items that assess the perceived availability of social support.
Interpersonal support at baseline | Baseline
  Measured using the Interpersonal Support Evaluation Checklist - 6 (ISEL-6). ISEL-6 is derived from the long form of the ISEL and contains 6 items that assess the perceived availability of social support.
Change in anti-HIV medication adherence | Through study completion, an average of 1 year
  Measured using the brief adherence self-report questionnaire. This questionnaire asks participants how much of their anti-HIV medications they have taken over the past month (0 to 100%).
Anti-HIV medication adherence at baseline | Baseline
  Measured using the brief adherence self-report questionnaire. This questionnaire asks participants how much of their anti-HIV medications they have taken over the past month (0 to 100%).
Change in frailty | Through study completion, an average of 1 year
  Measured using the Frailty Index Elders (FIFE). FIFE is a 10-item instrument with scores ranging from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty.
Frailty at baseline | Baseline
  Measured using the Frailty Index Elders (FIFE). FIFE is a 10-item instrument with scores ranging from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty.

SECONDARY OUTCOMES:
Demographic characteristics | Baseline, and once a year through study completion.
  Demographic characteristics including, but not limited to, age, sex, race, body weight, income, and education will be evaluated as potential predictors of inter- and intra-participant variability for patient-reported outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Mazonson & Santas Inc, Larkspur, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazonson P, Berko J, Lowman E, Gilliam B, Nwafor T, Clark A, Zolopa A. Number of Sexual Partners and Patient-Reported Outcomes Among Men Age 50+ with HIV. AIDS Res Hum Retroviruses. 2023 Oct;39(10):541-546. doi: 10.1089/aid.2023.0004. Epub 2023 Jun 28. PMID 37379478

DOCUMENTS (1):
  • Informed Consent Form (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04311554/ICF_000.pdf